CLINICAL TRIAL: NCT03432468
Title: Effect of Fully Blocking Type 1 Angiotensin Receptor on Blood Pressure, Cardiac Structure, Cardiac Function and Cognitive Function in Postmenopausal Hypertensive Women
Brief Title: Effect of Fully Blocking Type 1 Angiotensin Receptor on Target Organ Damage of Postmenopausal Hypertensive Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LanZhou University (Other)
Responsible Party: Principal Investigator, Jing Yu, Principal Investigator, LanZhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LanZhouU
Record Dates: First submitted 2018-01-19; First posted 2018-02-14 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-01

CONDITIONS: Hypertension
Keywords: Hypertension; Left Ventricular Hypertrophy; Women
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular | interventions — Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- postmenopausal hypertensive women (Active Comparator)
  Interventions: Drug: Valsartan 1; Drug: Valsartan 80 mg
- age-matched hypertensive male patients (Placebo Comparator)
  Interventions: Drug: Valsartan 1

INTERVENTIONS:
Drug: Valsartan 1 — the high dose of valsartan
Drug: Valsartan 80 mg — a single dose of valsartan
  Arms: postmenopausal hypertensive women

SUMMARY:
This study compared the improvements of blood pressure levels, left ventricular hypertrophy, left ventricular diastolic function, vascular function and cognitive function between postmenopausal hypertensive women and age-matched hypertensive male patients through the evaluation of the effects of fully blocked AT1 receptor by valsartan. Additionally, the differences of the above indexes between the patients who were fully blocked AT1 receptor by valsartan and the patients who were treated with a single dose of valsartan treatment were assessed, so as to provide theory basis for clinical treatment of postmenopausal hypertensive women.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypertension
* Women are all postmenopausal
* Must provide written informed consent

Exclusion Criteria:

* Secondary hypertension
* Coronary disease
* Heart failure
* Arterial fibrillation
* Previous myocardial infarction
* Previous stroke
* Malignant disease
* Kidney failure
* Liver failure
* Neoplastic disease
* Severe neurological diseases
* Severe metabolic or organic decompensation
* Refuse to sign the informed consent form

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Relative indexes of myocardial remodeling | Change from Baseline left ventricular mass index at 6 months.
  Cardiac structure (left ventricular mass index in grams for square meter) measurement.
Relative indexes of myocardial remodeling | Change from Baseline left ventricular mass index at 12 months.
  Cardiac structure (left ventricular mass index in grams for square meter) measurement.
Ambulatory blood pressure monitoring | Change from Baseline ABPM at 6 months.
  Non-invasive ambulatory blood pressure monitoring (ABPM) was performed for every enrolled patient with an ABPM equipment.
Ambulatory blood pressure monitoring | Change from Baseline ABPM at 12 months.
  Non-invasive ambulatory blood pressure monitoring (ABPM) was performed for every enrolled patient with an ABPM equipment.
Sexual hormones | Baseline sexual hormones.
  Blood samples used to analyze the levels of sexual hormones were collected between morning 8:00 and 9:00 after an overnight fast. The sexual hormones which include prolactin (PRL) and progesterone (P) units on nanogram per millilitre, luteinizing hormone (LH) and follicle-stimulating hormone (FSH) units on millionInternationalUnits per millilitre, testosterone (T) in nanogram per deciliter, estradiol (E2) in picogram per millilitre.

IPD SHARING:
Plan to Share IPD: Undecided